CLINICAL TRIAL: NCT04875377
Title: Iodine From Seaweed - a Randomised Controlled Trial of Food Versus Supplementation in Women With Marginal Habitual Iodine Intake
Brief Title: Seaweed Iodine Delivered Via Food or Supplementation
Acronym: INNOVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Emilie Combet, Principal Investigator, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 133109
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Iodine Deficiency
Keywords: iodine; seaweed; supplementation; reformulation; food matrix; thyroid function

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: Masking of pizzas was achieved by the use of pizzas with identical appearance and taste.
  Iodine and control supplements were also identical in appearance. Both pizzas and supplements were provided to investigators already masked. Pizzas labelled X and Y. Supplements labelled A and B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reformulated pizza (Experimental): Participants must consume a nutritionally balanced pizza reformulated with seaweed (Ascophyllum nodosum) as an ingredient 3 times a week for 24 weeks
  Interventions: Dietary Supplement: Reformulated pizza
- Control pizza (Placebo Comparator): Participants must consume a nutritionally balanced pizza without seaweed, 3 times a week for 24 weeks
  Interventions: Dietary Supplement: Control pizza
- Seaweed capsule (Experimental): Participants must consume a capsule containing powdered Ascophyllum nodosum 3 times a week for 24 weeks
  Interventions: Dietary Supplement: Seaweed capsule
- Control capsule (Placebo Comparator): Participants must consume an empty capsule 3 times a week for 24 weeks
  Interventions: Dietary Supplement: Control capsule

INTERVENTIONS:
Dietary Supplement: Reformulated pizza — Reformulated food with 400ug of iodine per meal, three times per week (to achieve 122% of weekly recommended intakes - average 140ug/day).
  Arms: Reformulated pizza
Dietary Supplement: Control pizza — Control (placebo) meal to consume thrice weekly (no iodine supplementation).
  Arms: Control pizza
Dietary Supplement: Seaweed capsule — Capsules containing seaweed extract, the iodine-rich ingredient in the reformulated pizza, 400ug iodine per capsule, to be consumed three times per week (122% of weekly recommended intake).
  Arms: Seaweed capsule
Dietary Supplement: Control capsule — Empty capsules (placebo)
  Arms: Control capsule

SUMMARY:
In this project, the investigators propose an intervention design testing the efficacy of a food reformulated with seaweed as an ingredient in meal, capsules against placebo and no intervention controls. The randomised control trial (supplementation) will last 24 weeks. The aim is to study the effect of the food matrix on variables associated with iodine nutrition: iodine status and thyroid function.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled trial conducted in Glasgow, United Kingdom. Inclusion criteria are as follows: healthy premenopausal women aged 18 - 60 years who would remain a resident in Glasgow for 24 weeks; who were self-reported low iodine consumers consuming milk less than once per day and non-oily fish less than once per week. Those with a history of thyroid dysfunction, taking medications other than the contraceptive pill or smoking, as well as pregnant or lactating women and those planning to conceive, were excluded. Those taking dietary supplements containing iodine would also excluded and there was no restriction related to body mass index (BMI).

Participants are recruited via social media and advertisements displayed around the Greater Glasgow area. Interested parties are screened and, if eligible, invited to a 30-minute appointment at which participants were randomly assigned through a web-based randomisation service to one of four groups after consent is obtained; reformulated pizza, control pizza, iodine capsules, or placebo capsules. During this initial meeting anthropometric measurements, blood pressure and a venous blood sample are collected, and participants are also asked to complete a sociodemographic questionnaire and an iodine specific food frequency questionnaire (FFQ). Participants are provided with instructions and equipment to record a 3-day estimated food diary and to collect 12 spot urine samples at different times of day over 2-7 days. Upon returning the spot urine samples, participants were given either the pizzas or supplements to begin the intervention. Participants are asked to consume one pizza or supplement three times a week for 24 weeks. Participants are asked to collect a further 10-12 sample spot urine samples at week 2 of the intervention. Participants are asked to attend another 30-minute appointment at 12 and 24 weeks in which baseline measurements are repeated along with a change to diet questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* self-reported healthy women
* aged 18 to 60
* pre-menopausal
* with no history of thyroid dysfunction
* without any known allergic reactions to foods
* not on medication that impact on absorption of nutrients from the gut
* not currently taking dietary / multivitamin supplements (must have discontinued usage 2 weeks prior the start of the study)

Exclusion Criteria:

* pregnancy
* lactation
* habitual consumption of seaweed-based products (>once per week), milk (>once per day), sea fish, non-oily, e.g. cod (>once per week)
* veganism (as food products contains cheese)
* Involvement in another research study where diet is restricted, modified, or dietary habits are studied.
* women who have reached menopause.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Change in urinary iodine concentration (UIC) | 0, 12 weeks
  Change in UIC assessed in pooled spot urine samples at 12 weeks, from baseline
Change in urinary iodine concentration (UIC) | 0, 24 weeks
  Change in UIC assessed in pooled spot urine samples at 24 weeks, from baseline

SECONDARY OUTCOMES:
Changes in body weight | 0, 12, 24 weeks
  Changes in body weight assessed from baseline at 12 and 24 weeks
Changes in body mass index | 0, 12, 24 weeks
  Changes in body mass index assessed from baseline at 12 and 24 weeks
Changes in waist circumference | 0, 12, 24 weeks
  Changes in waist circumference assessed from baseline at 12 and 24 weeks
Concentration of thyroid stimulating hormone | 0, 12, 24 weeks
  measured by immunoassay
Concentration of thyroglobulin | 0, 12, 24 weeks
  measured by immunoassay
Concentration of Free Triiodothyronine | 0, 12, 24 weeks
  measured by immunoassay
Concentration of Thyroxine | 0, 12, 24 weeks
  measured by immunoassay
Dietary iodine intake | 0, 12, 24 weeks
  estimated by food frequency questionnaire (FFQ)
Change in urinary iodine concentration (UIC) | 0, 2 weeks
  Change in UIC assessed in pooled spot urine samples at 2 weeks, from baseline

OTHER OUTCOMES:
concentration of triglycerides | 0, 12, 24 weeks
  measured in blood
concentration of total cholesterol | 0, 12, 24 weeks
  measured in blood
concentration of HDL/LDL cholesterol | 0, 12, 24 weeks
  measured in blood
glucose concentration | 0, 12, 24 weeks
  measured in blood

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Combet, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No